CLINICAL TRIAL: NCT06694454
Title: Phase I/II Study of Neoadjuvant Inhaled Azacytidine With Platinum-Based Chemotherapy and Durvalumab (MEDI4736) - a Combined Epigenetic-Immunotherapy (AZA-AEGEAN) Regimen for Operable Early-Stage Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Neoadjuvant Inhaled Azacytidine With Platinum-Based Chemotherapy and Durvalumab (MEDI4736) - a Combined Epigenetic-Immunotherapy (AZA-AEGEAN) Regimen for Operable Early-Stage Non-Small Cell Lung Cancer (NSCLC)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10001609; 001609-C
Record Dates: First submitted 2024-11-16; First posted 2024-11-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09-05

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); Carcinoma, Non-Small Cell Lung; Non-Small Cell Lung Carcinoma; Non Small Cell Lung Cancer; Non Small Cell Lung Carcinoma
Keywords: immune checkpoint inhibitor (CPI); pathologic complete response (pCR); aerosolized drug delivery; immunosuppressive tumor microenvironment (TME); reversible epigenetic mechanisms; DNA demethylating agents; nebulizer treatment; AZA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pathologic Complete Response | interventions — Azacitidine; Carboplatin; Paclitaxel; durvalumab; Cisplatin; Gemcitabine; Pemetrexed

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/ Phase I Dose Escalation (Experimental): Histology specific SOC platinum-based chemotherapy with durvalumab plus escalating/de-escalating doses of aerosolized azacytidine
  Interventions: Drug: azacytidine; Drug: carboplatin; Drug: paclitaxel; Drug: durvalumab; Drug: cisplatin; Drug: gemcitabine; Drug: pemetrexed
- 2/ Phase II Dose Expansion (Experimental): Histology specific SOC platinum-based chemotherapy with durvalumab plus RP2D of aerosolized azacytidine
  Interventions: Drug: azacytidine; Drug: carboplatin; Drug: paclitaxel; Drug: durvalumab; Drug: cisplatin; Drug: gemcitabine; Drug: pemetrexed

INTERVENTIONS:
Drug: azacytidine — Aerosolized azacytidine (AZA) via nebulizer on 3 consecutive days during the first week of every cycle (1 cycle=21 days), for a maximum (total) of 3 cycles.
  Azacytidine will be given at escalating doses in phase 1, and at the established RP2D in phase 2.
Drug: carboplatin — Carboplatin (intravenous/IV), area under the serum drug concentration-time curve (AUC)=5-6 mg/mL/min based on cancer histology administered on day 4 of every cycle (1 cycle=21 days), for a maximum (total) of 3 cycles.
Drug: paclitaxel — Paclitaxel (IV), 200 mg/m^2, is administered on day 4 of every cycle (1 cycle=21 days), for a maximum (total) of 3 cycles.
Drug: durvalumab — Durvalumab (IV) administered as a flat dose of 1500 mg on day 4 of every cycle (1 cycle=21 days), for a maximum (total) of 3 cycles.
Drug: cisplatin — Cisplatin (IV), 75 mg/m^2, administered on day 4 of every cycle (1 cycle=21 days), for a maximum (total) of 3 cycles.
Drug: gemcitabine — Gemcitabine (IV), 1,250 mg/m^2, administered on day 4 of every cycle (1 cycle=21 days), for a maximum (total) of 3 cycles.
Drug: pemetrexed — Pemetrexed (IV), 500 mg/m^2, administered on day 4 of every cycle (1 cycle=21 days), for a maximum (total) of 3 cycles.

SUMMARY:
Background:

Lung cancer is the leading cause of cancer-related death worldwide. Non-small cell lung cancer (NSCLC) is the most common type of lung cancer. Surgery to remove the tumors is the standard treatment for people diagnosed with early stages of NSCLC. Despite complete removal of these tumors, many recur (happen again). An FDA-approved drug combination to treat early-stage NSCLC prior to the surgery is durvalumab plus standard chemotherapy. The FDA approved infusion drug azacytidine [AZA] is used to treat several diseases because it can rapidly kill dividing cells (including cancer cells) but it is not approved for NSCLC. An inhaled (aerosolized) form of AZA is also not approved for NSCLC. However, researchers want to know if an inhaled version of AZA can help improve treatment of people with NSCLC because inhaled AZA goes directly into the lungs with limited absorption into the bloodstream.

Objective:

To find the safest and most effective dose of inhaled AZA in participants with early-stage non-small cell lung cancer (NSCLC) that can still be removed by surgery.

Eligibility:

Adults aged 18 and older with operable early-stage NSCLC. Participants will be required to also enroll in NIH protocol 06C0014 which allows for pre- and post-treatment biopsies and bloodwork to be obtained for additional research studies.

Design:

Participants will be screened. They will have a physical exam with blood tests. Their medical records will be reviewed. They will have imaging scans and tests of their heart and lung functions. Participants will be required to have a tissue sample (biopsy) taken of their tumor prior to receiving study drug and again during surgery after Cycle 3; airway tissue biopsies and collection of collect bronchial (lung) fluid may also be done.

Participants will receive the study treatment for 3 cycles. Each cycle is 21 days. They will need to come to the NIH Clinical Center (CC) on days 1-4 of Cycles 1-3.

AZA will be given as a drug mist that can be inhaled (like the type of mist in an asthma inhaler) using a nebulizer at the NIH Clinical Center (CC) for 3 days in a row (consecutive days) during the first week of each cycle. The participant will inhale the AZA drug mist for 20 to 30 minutes each time. Participants will also receive durvalumab and a specific 2-drug assigned chemotherapy by intravenous (IV) infusion on day 4 of each cycle.

Participants will have a follow-up visit 2 weeks after their last dose of study drugs. Then they will have planned surgery to remove the tumors.

Participants will have additional follow-up visits at the NIH CC about 1 and 3 months after the surgery, and then for every 3 months for up to 3 years.

...

DETAILED DESCRIPTION:
Background:

* Lung cancer is the leading cause of cancer-related mortality worldwide and accounted for nearly 160,000 deaths in 2023 in the US.
* Paradigm shifting results of immune checkpoint inhibitor (CPI) therapy in locally advanced, inoperable, and metastatic non-small cell lung cancer (NSCLC) have prompted clinical evaluation of these agents administered in the perioperative setting for patients with earlystage, operable disease.
* Pathologic complete responses (pCR) are observed in approximately 10% of early-stage NSCLC following CPI monotherapy and between 20-30% following platinum based chemotherapy and CPI treatment; as such most NSCLC are intrinsically resistant to immune checkpoint blockade.
* Many of the pathways that drive pulmonary carcinogenesis and render NSCLC resistant to immunotherapy are mediated by potentially reversible epigenetic mechanisms of which DNA methylation appears to be predominant.
* DNA demethylating agents such as azacytidine and decitabine can directly enhance the immunogenicity of lung cancer cells and ameliorate immunosuppression within the tumor microenvironment (TME).
* Poor bioavailability, as well as pharmacokinetic/pharmacodynamic limitations and systemic toxicities prevent optimal dosing of DNA demethylating agents for the treatment of solid tumors.
* One potential strategy to enhance the delivery of DNA demethylating agents to early-stage NSCLC while minimizing systemic toxicities is to administer these drugs by inhalation techniques.
* Preclinical studies have demonstrated that aerosolized AZA mediates epigenetic activation of tumor suppressor gene expression in orthotopic human NSCLC, and significantly prolongs the survival of mice bearing these xenografts without systemic toxicities.
* Conceivably, by simultaneously targeting lung cancer cells and their immunosuppressive TME, inhaled AZA may enhance the efficacy of chemo-immunotherapy for early-stage NSCLC.

Objectives:

* Phase I:

  --To determine the maximum tolerated dose (MTD) and the recommended phase II dose (RP2D) of neoadjuvant aerosolized AZA in participants with operable early-stage NSCLC treated with standard of care (SOC) platinum-based chemotherapy and Durvalumab.
* Phase II:

  * To determine the frequency of pathologic complete responses (pCR) in participants receiving aerosolized AZA, durvalumab, and SOC platinum-based chemotherapy as induction therapy for early-stage NSCLC.

Eligibility Criteria:

* Stage IB-IIIA NSCLC irrespective of programmed death-ligand 1 (PD-L1) expression status.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* No prior therapy for NSCLC.
* Disease that can be safely accessed via bronchoscopic, thoracoscopic, or percutaneous biopsy, and participant willingness to undergo tumor biopsy before treatment (all participants) and bronchoscopic evaluation for PK analysis during treatment (Phase I only).
* Willing to undergo tumor resection per standard of care (SOC) guidelines following induction therapy.
* Age >=18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of <=1.
* Adequate organ and marrow function.

Design:

* Eligible participants will receive aerosolized AZA via AeroEclipse(R) II Breath Actuated nebulizer on three consecutive days (i.e., days 1, 2, 3) of a 21-day cycle for 3 cycles. Platinumdoublet chemotherapy using SOC guidelines and durvalumab will be administered on day 4 of each cycle.
* Anatomic resection [lobectomy/segmentectomy/pneumonectomy with mediastinal lymph node dissection (MLND)] will be performed within 3 weeks following completion of neoadjuvant therapy regimen.
* The dose of AZA will be escalated using a 3+3 design with no intra-patient dose escalation (45 - 75 mg/m^2/inhalation) to maximize intra-tumoral DNA methyltransferase (DNMT) 1 depletion while avoiding dose-limiting pulmonary or systemic toxicities attributable to this agent during the three cycles of therapy.
* Once the RP2D of aerosolized AZA has been defined either by toxicity or feasibility, that cohort will be expanded to a total of 17 participants to determine pathologic complete response rates at the RP2D using a Simon optimal design for phase II trials.
* If 4 or more of 17 participants treated at the RP2D experience pCR, an additional 20 evaluable participants will be accrued (2nd stage).
* Pharmacokinetic (PK) / pharmacodynamic (PD) effects as well as DNMT, CTA, and immune-related gene expression levels in tumor tissues may be evaluated.
* Additional studies will be performed to examine if the treatment regimen alters DNA methylation and cytokine levels and modulates the phenotypes of immune cells in pulmonary lavage fluids.
* Up to 52 participants may receive study intervention on this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologically or cytologically confirmed, resectable per standard of care stage IB-IIIA non-small cell lung cancer (NSCLC) irrespective of programmed death-ligand 1 (PD-L1) expression. Note: Confirmation is required by NCI Laboratory of Pathology (LP).
* Willingness to undergo tumor resection surgery per standard of care (SOC) guidelines following induction therapy (platinum chemotherapy and durvalumab).
* Participants must have disease that can be safely accessed via bronchoscopic, thoracoscopic, or percutaneous biopsy techniques, and be willing to undergo tumor biopsy before treatment.
* No prior therapy for the NSCLC.
* Measurable disease per RECIST 1.1
* Age >= 18 years.
* Body weight > 30kg.
* ECOG Performance Status <= 1
* Participants must have adequate pulmonary reserve evidenced by predicted post-op FEV1 and adjusted DLCO >= 40% at screening.
* Participants must have pCO2 <= 45 and pO2 >=60 on room air by arterial blood gas (ABG) if O2 sat by pulse oximetry is<= 92% on room air at screening.
* Adequate organ and marrow function as defined below:

  * Leukocytes >3,000/microL
  * Absolute neutrophil count >1,500/microL (without transfusion or cytokine support)
  * Absolute lymphocyte count > 800/microL
  * Platelets >100,000/microL
  * Hemoglobin >= 9.0 g/dL
  * Prothrombin time (PT) no more than 2 seconds above the upper limit of normal (ULN)
  * Total bilirubin OR Direct bilirubin < 1.5 X institutional upper limit of normal OR <= ULN for participants with total bilirubin >= 1.5 ULN
  * Aspartate aminotransferase (AST) / Alanine aminotransferase (ALT) < 2.5 X institutional ULN
  * Serum albumin >= 2.0 mg/dL
  * Creatinine OR Creatinine clearance (eGFR) <= 1.6 mg/ml OR >60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal
* Individuals of child-bearing potential (IOCBP) must agree to use a highly effective method of contraception (hormonal, intrauterine device (IUD), surgical sterilization, abstinence) for the duration of the study treatment and up to 6 months after the last dose of the study drug(s). Note: participants who have cisplatin as part of SOC chemo must agree to use a highly effective method of contraception for 14 months.

Individuals able to father a child must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) for the duration of the study treatment and up to 3 months after the last dose of the study drug(s). Note: participants who have cisplatin as part of SOC chemo must agree to use an effective method of contraception for 11 months. We also will recommend these individuals with partners of childbearing potential to ask partners to be on highly effective birth control (hormonal, intrauterine device (IUD), surgical sterilization).

* Breastfeeding participants must be willing to discontinue breastfeeding from study treatment initiation through 3 months after the last dose of the study drug(s).
* Participants with history of human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness are included if on appropriate antiretroviral therapy with HIV viral load <400 copies/mL.
* Participants must agree to not donate blood from the study entry and up to 3 months after the last dose of the study drug(s).
* Participants must be co-enrolled in protocol 06C0014: Prospective Evaluation of Genetic and Epigenetic Alterations in Patients with Thoracic Malignancies .
* The ability of a participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Medically inoperable because of clinical co-morbidities.
* Participants with T4 tumors invading the diaphragm, mediastinum, carina, trachea, esophagus, heart, great vessels, recurrent laryngeal nerve, or vertebral body.
* Participants who experienced serious immune adverse events that required discontinuation of immune checkpoint inhibitor therapy for a prior non-NSCLC malignancy.
* History of known EGFR or ALK alterations in the tumor.
* History of active autoimmune disease including colitis, nephritis, hypophysitis, or neuropathy, with the exceptions of:

  --Diabetes type I, vitiligo, alopecia, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment.
* History of pneumonitis or interstitial lung disease.
* Clinically significant cardiovascular/cerebrovascular disease as follows:

  * cerebral vascular accident/stroke (within 6 months prior to study treatment initiation)
  * myocardial infarction (within 6 months prior to study treatment initiation)
  * unstable angina, congestive heart failure (New York Heart Association Classification Class >= II, https://manual.jointcommission.org/releases/TJC2016A/DataElem0439.html#:~:text=Class%20II%20%2D%20Mild%20symptoms%20(mild,Class%20IV%20%2D%20Severe%20limitations), serious cardiac arrhythmia, clinically significant bleeding or clinically significant pulmonary embolism at screening.
* Active Hepatitis A (HAV), Hepatitis B (HBV) (HbsAg reactive), or Hepatitis C (HCV) (HCV RNA [qualitative] is detected) at screening.
* Other active infections requiring systemic therapy at screening.
* Positive beta human chorionic gonadotropin (beta-HCG) serum or urine pregnancy test performed in females of childbearing potential at screening.
* Systemic corticosteroids at doses above physiologic levels (> 10 mg of prednisone or equivalent per day), or inhaled corticosteroids within 14 days before study treatment initiation. Administration of steroids through a route known to result in a minimal systemic exposure (i.e., topical, intro-ocular, or intra-articular) is allowed.
* Major surgical procedure within 28 days prior to the study treatment initiation. Note: Local surgery of isolated lesions for palliative intent is acceptable provided other site(s) of disease is available for response assessment.
* History of allogenic organ transplantation.
* History of another primary malignancy except for malignancy treated with curative intent and with no known active disease >= 5 years before the study treatment initiation.
* Administration of live attenuated vaccines within 30 days prior to study treatment initiation. Note: Administration of inactivated vaccines (e.g., inactivated influenza vaccines) is permitted before or during the study.
* Administration of investigational drug on other clinical trial within 14 days prior to study treatment initiation.
* History of hypersensitivity to Mannitol.
* Herbal and natural remedies that may have immune-modulating effects within 7 days prior to study treatment initiation.
* Uncontrolled intercurrent illness evaluated by history and physical exam or situation that would limit compliance with study requirements.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase I: To determine the maximum tolerated dose (MTD) and the recommended phase II dose (RP2D) of neoadjuvant aerosolized AZA in participants with operable early-stage NSCLC treated with standard of care (SOC) platinum-based chemotherapy and du... | starts at initiation of study drug, though end of DLT period
  DLTs noted at each dose level will be reported.
Phase II: To determine the frequency of pathologic complete responses (pCR) in participants receiving aerosolized AZA, durvalumab, and SOC platinum-based chemotherapy as induction therapy for early-stage NSCLC | baseline (pre-treatment biopsy), and at the time of SOC surgery post-cycle 3
  Pathologic complete responses (pCR) is defined as no viable cancer cells in samples collected on histopathologic assessment. Fraction of evaluable participants who experience a pCR will be determined and reported along with 80% and 95% two-sided confidence intervals.

SECONDARY OUTCOMES:
To evaluate pharmacokinetics | All participants: Cycle 1, Day 1 or 2, and Cycle 3, Day 1 or 2. Participants with MTD treatment: Cycle 1, Day 1 or 2, and Cycle 2, Day 1 or 2, and Cycle 3, Day 1 or 2.
  Pharmacokinetic endpoints will be reported using descriptive statistics.
To evaluate safety of the combination of AZA and chemo-durvalumab in participants with operable early-stage NSCLC | starts at initiation of study drug, through 64 days after the last study drug administration
  Safety of the agents will be assessed by determining the grade of adverse events noted in each participant and reporting the fraction with Grade 3 and Grade 4 adverse events. Safety data will be presented in a summary. The safety data will consist of the reporting of all adverse events, and may also include reporting vital signs, physical examination data, and laboratory safety data.
To evaluate event-free survival (EFS) | baseline, Day 64 (treatment evaluation), then post-surgical 1 month, 3 months, and every 3 months thereafter until disease progression, until up to 3 years from the treatment initiation
  Event-free survival (EFS) at three years post treatment will be determined as the duration of time from start of treatment to time of disease recurrence or appearance of new primary cancer, whichever occurs first as appropriate using the Kaplan-Meier method and reported along with a 95% confidence interval, separately for phase I and II. The median EFS will also be reported along with a 95% confidence interval.
To evaluate objective response (complete response [CR] + partial response [PR]) and stable disease [SD] per RECIST 1.1 | baseline, and at Day 64 (treatment evaluation)
  The objective response rate will be based on CR+PR and the disease stabilization rate (SD) and reported separately in phase I and II along with a 95% confidence interval for each.
To evaluate major pathologic response (MPR) rate | baseline (pre-treatment biopsy), and at the time of SOC surgery post-cycle 3
  MPR rate is defined as <10% viable cancer cells in samples collected per histopathologic assessment. The objective response rate based on the MPR rate will be reported separately in phase I and II along with a 95% confidence interval for each.

CONTACTS AND LOCATIONS:
Overall Officials: David S Schrump, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing. This study will comply with the NIH Genomic Data Sharing (GDS) Policy, which applies to all new and ongoing NIH IRP-funded research, as of January 25, 2015, that generates large-scale human or non-human genomic data, as well as the use of these data for subsequent research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study will be shared after the completion of the primary endpoint per the data management sharing plan.
Access Criteria: Data from this study may be requested by contacting the PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001609-C.html